CLINICAL TRIAL: NCT01607710
Title: Locating Regions of Interest in Generalized Anxiety Disorder Using Function Magnetic Resonance Imaging (fMRI)
Acronym: fMRI
Status: Completed | Type: Observational
Sponsor: Hartford Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: DIEF003523.2
Record Dates: First submitted 2012-05-25; First posted 2012-05-30 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2013-03

CONDITIONS: Generalized Anxiety Disorder
Keywords: fMRI; Generalized Anxiety Disorder
MeSH Terms: conditions — Generalized Anxiety Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Generalized Anxiety Disorder: The group of participants diagnosed with generalized anxiety disorder.
- Nonclinical Control Group: The comparison group of participants with no psychiatric diagnoses.

SUMMARY:
The investigators are seeking to locate the brain regions of interest in generalized anxiety disorder (GAD) using both structural (sMRI) and functional magnetic resonance imaging (fMRI). The MRI will be used to measure changes in blood flow in the brain while at rest and while completing tasks designed to elicit symptoms of anxiety. Results from a nonclinical control group and a GAD group will be compared to determine whether they exhibit different areas of brain activity during the tasks.

DETAILED DESCRIPTION:
20 healthy controls and 20 participants with GAD will be recruited. Each participant will undergo an MRI session that will last approximately 2 hours. The structural MRI will be used when the participant is at rest. During the functional MRI (fMRI), a computer screen inside the scanner will display four tasks the participant must complete: (1)Gambling Task, (2)Risk & Ambiguity Task, (3)Reading Emotion from the Eyes (REE) Task, and (4)Emotional Counting Task.

ELIGIBILITY:
Generalized Anxiety Disorder(GAD)Group:

Inclusion Criteria:

* Clinical diagnosis of Generalized Anxiety Disorder
* Hamilton Anxiety Rating Scale score of 18 or higher
* Hamilton Rating Scale for Depression score of 17 or less
* Fluency in English
* Capacity to understand the nature of the study and willingness to sign informed consent for

Exclusion Criteria:

* History of epilepsy or head trauma (Loss of consciousness>5 minutes) with the past 6 months
* Lifetime history of increased intracranial pressure, seizure disorder, stroke, brain tumor, multiple sclerosis or brain surgery
* A review of patient medications by the study physician indicates an increased risk of seizure
* An active autoimmune, endocrine, viral, or vascular disorder affecting the brain; any unstable cardiac disease; hypertension; or severe renal or liver insufficiency
* Substance use disorder or posttraumatic stress disorder (PTSD) within the past 6 months
* Lifetime bipolar disorder, obsessive-compulsive disorder (OCD), psychotic disorder, mental retardation, or pervasive development disorder
* Any psychotic features, including dementia or delirium
* Medication change within past 3 months
* Current serious suicidal or homicidal ideation, and/or serious suicidal attempt within past 6 months
* Serious, unstable, or terminal medical condition or clinically judged too psychiatrically unstable to participate in the study
* Any contraindication for participation in MRI scan

Nonclinical Control Group:

Inclusion Criteria:

* Absence of any psychiatric diagnosis

Exclusion Criteria:

* History of epilepsy or head trauma (Loss of Consciousness>5 minutes) with the past 6 months
* Lifetime history of increased intracranial pressure, seizure disorder, stroke, brain tumor, multiple sclerosis or brain surgery
* A review of patient medications by the study physician indicates an increased risk of seizure
* An active autoimmune, endocrine, viral, or vascular disorder affecting the brain; any unstable cardiac disease; hypertension; or severe renal or liver insufficiency
* Substance use disorder or PTSD within the past 6 months
* Lifetime bipolar disorder, OCD, psychotic disorder, mental retardation, or pervasive development disorder
* Any psychotic features, including dementia or delirium
* Medication change within past 3 months
* Current serious suicidal or homicidal ideation, and/or serious suicidal attempt within past 6 months
* Serious, unstable, or terminal medical condition or clinically judged too psychiatrically unstable to participate in the study
* Any contraindication for participation in MRI scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Residents of the Greater Hartford Connecticut area.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2012-07; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Brain activation while undergoing the fMRI | Throughout the fMRI
  Main effects for each condition will be calculated to elucidate brain activations relevant to the tasks. Random effect 2 sample t-tests will assess group differences (i.e., GAD patients vs. healthy controls) to identify regions that demonstrate hyperactivation in patients.

CONTACTS AND LOCATIONS:
Overall Officials: Gretchen J Diefenbach, Ph.D., Principal Investigator — Hartford Hospital
Locations (1):
- Hartford Hospital, Hartford, Connecticut, United States